CLINICAL TRIAL: NCT05425966
Title: Adapting a Remote Training for Mexican School Clinicians Delivering Evidence-Based Intervention for ADHD and ODD
Brief Title: Adapting a Web-Based Professional Development for Mexican School Mental Health Providers Delivering Evidence-Based Intervention for ADHD and ODD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLSRFUERTE; R21MH124066 (NIH)
Record Dates: First submitted 2022-06-15; First posted 2022-06-21 (Actual); Results first posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: ADHD; Oppositional Defiant Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Oppositional Defiant Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CLS-R-FUERTE (Experimental): Active program participation in: a remote school clinician training and comprehensive psychosocial intervention designed to improve attention and behavior in Mexican school-aged youth (grades 1-5). via school clinician training by a clinical research team to lead parent skill groups, child skill groups, and teacher consultation in a behavioral classroom management system.
  Interventions: Behavioral: CLS-R-FUERTE

INTERVENTIONS:
Behavioral: CLS-R-FUERTE — The CLS-R-FUERTE program is a remote school clinician training and comprehensive psychosocial intervention designed to improve attention and behavior in Mexican school-aged youth (grades 1-5). It contains the same evidence-based service components to improve youth attention/behavior as the in-person CLS-FUERTE program; specifically, it features school clinician training by a clinical research team to lead parent skill groups, child skill groups, and teacher consultation in a behavioral classroom management system.

SUMMARY:
Neurodevelopmental disorders of inattention and disruptive behavior, such as Attention-Deficit/ Hyperactivity Disorder (ADHD) and Oppositional Defiant Disorder (ODD), are among the most common youth mental health conditions across cultures. An efficacious and feasible solution to improving affected youth's ADHD/ODD is training existing school clinicians to deliver evidence-based intervention with fidelity. Despite initial promising results of training school clinicians to treat ADHD/ODD in settings suffering from high unmet need, such as Mexico, scalability is limited by a lack of researchers with capacity to train, monitor, and evaluate school clinicians in such efforts on a large scale. Thus, there is a need to develop more feasible interventions and training programs for school clinicians, as well as create a system with capacity for scalable training and evaluation, to combat the widespread impact ofADHD/ODD worldwide. Converting interventions and school clinician professional development programs for fully-remote delivery allows for more flexibility, accessibility, affordability, scalability, and promise for ongoing consultation than in-person options. Supporting scalable training for school clinicians could address a significant public health concern in Mexico, as only 14% of Mexican youth with mental health disorders receive treatment and less than half of those treated receive more than minimally adequate care. The study team is uniquely suited for this effort, given that they developed the only known school-homeADHD/ODD evidence-based intervention in Latin America-and-have developed a web-based training for U.S. school clinicians with promising preliminary results. The study team's prior studies and high levels of unmet need make Mexico an ideal location for this proposal; however, lessons learned could be used to expand scalable school clinician training for evidence-based intervention in other settings and/or for other disorders. Thus, this study focuses on conducting an open-trial of the fully-remote program and make iterative changes. It is predicted that: H1) school clinicians trained remotely will be satisfied and show improved evidence-based practice skills; H2)families and teachers participating remotely will be satisfied and youth will show improved ADHD/ODD; H3) observation/feedback from a 3-school open-trial will guide iterative changes to the remote program.

ELIGIBILITY:
Inclusion Criteria:

* Students meeting the following criteria are eligible:

  * at least six inattention symptoms and/or six hyperactive/impulsive symptoms endorsed by parent or teacher as occurring often or very often,
  * at least one area of impairment rated as concerning by both parent and teacher, and
  * a parent and teacher agreeing to participate.
  * Students taking medication are eligible as long as regimens were stable.
* Parents and teachers and school clinicians of participating are eligible to participate.

Exclusion Criteria:

All Participants: Anyone who does not speak and read Spanish will be excluded, given that all informed consent, measurement, and activity procedures will be conducted in Spanish.

Child Participants

* Children taking medication will be eligible for screening after the child has been on a stable medication regimen for at least one month (to minimize chance that treatment effects are due to medication and not the proposed program).
* Presence of conditions that are incompatible with this study's treatment.
* severe visual or hearing impairment,
* severe language delay,
* psychosis,
* Child does not read or speak Spanish (inability to complete assessment measures or participate in group treatments).
* Child is in an all-day special education classroom. Children in these classrooms are frequently receiving intensive behavior modification programs and assistance such that the teacher consultation component would be expected to require modification for use in these settings.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lauren M Haack, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants who enrolled in the study were assigned to the CLS-R-FUERTE active treatment group and were included in the study.
Period: Overall Study
Arm/Group | CLS-R-FUERTE
Started | 67
Completed | 67
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | CLS-R-FUERTE
Number analyzed (Participants) | 67
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 23
  Between 18 and 65 years | 44
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] — Age collected for students in the study Population: Age was collected for the youth in the study
  years
    number analyzed (Participants) | 23
    (all) | 8.04 [6 to 11]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 67
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 67
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Mexico | 67
ADHD Presentation [Count of Participants; unit: Participants] — Population: ADHD presentation collected for students in the study
  Participants
    number analyzed (Participants) | 23
    Inattentive Profile | 9
    Combined Profile | 14
ODD Presentation [Count of Participants; unit: Participants] — Population: ODD presentation collected for students in the study
  Participants
    number analyzed (Participants) | 23
    (all) | 10
On medication % [Count of Participants; unit: Participants] — Population: collected for students in the study
  Participants
    number analyzed (Participants) | 23
    (all) | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Child Symptom Inventory-4 (CSI-4) Parent Checklist ADHD Combined Type Symptom Severity Score
Description: Parents will assess ADHD symptoms using the CSI-4. The CSI-4: Parent Checklist contains 18 symptoms for ADHD, Combined type (ADHD:C; 18 items). Each symptom is rated on a 4-point scale (0= never to 3= very often). The average of ADHD:C scores range from zero to four, with higher scores indicating more severe symptoms.
Time Frame: Baseline and post treatment (8 weeks)
Population: The 23 participants who were students were analyzed within this outcome measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CLS-R-FUERTE
Number analyzed (Participants) | 23
score on a scale | 0.82 (0.52)

2. Primary Outcome: Change in Child Symptom Inventory-4 (CSI-4) Teacher Checklist ADHD Combined Type Symptom Severity Score
Description: Teachers will assess ADHD symptoms using the CSI-4. The CSI-4: Teacher Checklist contains 18 symptoms for ADHD, Combined type (ADHD:C; 18 items). Each symptom is rated on a 4-point scale (0= never to 3= very often). The average of ADHD:C scores range from zero to four, with higher scores indicating more severe symptoms.
Time Frame: Baseline and post treatment (8 weeks)
Population: The 23 participants who were students were the target to be analyzed within this outcome measure data; there was missing teacher-report student outcome for 2 students; thus, the 21 participants who were students and had teacher-report outcome data were analyzed within this outcome measure data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CLS-R-FUERTE
Number analyzed (Participants) | 21
score on a scale | 0.68 (0.47)

3. Primary Outcome: Change in Child Symptom Inventory-4 (CSI-4) Parent Checklist (Oppositional Defiant Disorder) ODD Symptom Severity Score
Description: Parents will assess ODD symptoms using the CSI-4. The CSI-4: Parent Checklist contains 9 symptoms of ODD. Each symptom is rated on a 4-point scale (0= never to 3= very often). The average ODD scores range from zero to four, with higher scores indicating more severe symptoms.
Time Frame: Baseline and post treatment (8 weeks)
Population: The 23 participants who were students were analyzed within this outcome measure data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CLS-R-FUERTE
Number analyzed (Participants) | 23
score on a scale | 0.54 (0.62)

4. Primary Outcome: Change in Child Symptom Inventory-4 (CSI-4) Teacher Checklist (Oppositional Defiant Disorder) ODD Symptom Severity Score
Description: Teachers will assess ODD symptoms using the CSI-4. The CSI-4: Teacher Checklist contains 9 symptoms of ODD. Each symptom is rated on a 4-point scale (0= never to 3= very often). The average ODD scores range from zero to four, with higher scores indicating more severe symptoms.
Time Frame: Baseline and post treatment (8 weeks)
Population: The 23 participants who were students were the target to be analyzed within this outcome measure data; there was missing teacher-report student outcome for 4 students; thus, the 19 participants who were students and had teacher-report outcome data were analyzed within this outcome measure data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CLS-R-FUERTE
Number analyzed (Participants) | 19
score on a scale | 0.43 (0.55)

5. Primary Outcome: Change Impairment Rating Scale (IRS) Parent Questionnaire Overall Severity Score
Description: Parents will assess impairment using the IRS. The IRS Teacher Questionnaire contains 8 items of functional impairment (i.e., academic and peer relations). Each item is rated on a 7-point scale (1= no problem; does not need treatment/services to 7= extreme impairment; definitely needs treatment/services). The average of all IRS scores range from one to seven, with higher scores indicating more severe impairment.
Time Frame: Baseline and post treatment (8 weeks)
Population: The 23 participants who were students were analyzed within this outcome measure data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CLS-R-FUERTE
Number analyzed (Participants) | 23
score on a scale | 1.82 (1.15)

6. Primary Outcome: Change Impairment Rating Scale (IRS) Teacher Questionnaire Overall Severity Score
Description: Teachers will assess impairment using the IRS. The IRS Teacher Questionnaire contains 8 items of functional impairment (i.e., academic and peer relations). Each item is rated on a 7-point scale (1= no problem; does not need treatment/services to 7= extreme impairment; definitely needs treatment/services). The average of all IRS scores range from one to seven, with higher scores indicating more severe impairment.
Time Frame: Baseline and post treatment (8 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CLS-R-FUERTE
Number analyzed (Participants) | 21
score on a scale | 2.25 (1.23)

ADVERSE EVENTS:
Time Frame: 10 months
Arm/Group | CLS-R-FUERTE
All-Cause Mortality (participants affected / at risk) | 0/67
Serious Adverse Events (participants affected / at risk) | 0/67
Other Adverse Events (participants affected / at risk) | 0/67

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-08-22): https://cdn.clinicaltrials.gov/large-docs/66/NCT05425966/Prot_SAP_000.pdf
  • Informed Consent Form (2022-08-22): https://cdn.clinicaltrials.gov/large-docs/66/NCT05425966/ICF_001.pdf